CLINICAL TRIAL: NCT02342340
Title: A Blinded, Randomized, Controlled Study to Examine the Bioavailability of Compounds From Different Bean Varieties in Healthy Individuals.
Brief Title: Bioavailability of Compounds From Different Bean Varieties in Healthy Individuals.
Acronym: BBB-2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Peter Zahradka (Other)
Collaborators: Manitoba Pulse Growers (Other)
Responsible Party: Sponsor-Investigator, Dr. Peter Zahradka, Principal Investigator and Professor, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: B2014:122
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Beans, Lentils, Bioavailability, Phytochemical Absorption
MeSH Terms: interventions — Cooking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Navy Beans (cooked) (Active Comparator): At one of the six visits, participants will consume a ¾ cup of cooked navy beans. Participants will be provided with 100 ml of water with the food, and will be allowed to drink water whenever necessary during the 6 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 6 visits have been completed.
  Interventions: Other: Navy Beans (cooked)
- Red Kidney Beans (cooked) (Active Comparator): At one of the six visits, participants will consume a ¾ cup of cooked red kidney beans. Participants will be provided with 100 ml of water with the food, and will be allowed to drink water whenever necessary during the 6 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 6 visits have been completed.
  Interventions: Other: Red Kidney Beans (cooked)
- Pinto Beans (cooked) (Active Comparator): At one of the six visits, participants will consume a ¾ cup of cooked pinto beans. Participants will be provided with 100 ml of water with the food, and will be allowed to drink water whenever necessary during the 6 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 6 visits have been completed.
  Interventions: Other: Pinto Beans (cooked
- Black Beans (cooked) (Active Comparator): At one of the six visits, participants will consume a ¾ cup of cooked navy beans. Participants will be provided with 100 ml of water with the food, and will be allowed to drink water whenever necessary during the 6 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 6 visits have been completed.
  Interventions: Other: Black Beans (cooked)
- Lentils (cooked) (Active Comparator): At one of the six visits, participants will consume a ¾ cup of cooked lentils. Participants will be provided with 100 ml of water with the food, and will be allowed to drink water whenever necessary during the 6 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 6 visits have been completed.
  Interventions: Other: Lentils (cooked)
- White Rice (cooked) (Placebo Comparator): At one of the six visits, participants will consume a ¾ cup of cooked white rice. Participants will be provided with 100 ml of water with the food, and will be allowed to drink water whenever necessary during the 6 hour test period. The participants will not be blinded to the order and the type of food product they receive at a visit, however, the samples will be assigned a number to ensure the analytical team is blinded to the test product until the end of the study. Should the need to re-administer a test product arise, the participant will receive the test product from the same treatment number again at an extra visit after the original 6 visits have been completed.
  Interventions: Other: White Rice

INTERVENTIONS:
Other: Navy Beans (cooked) — One time consumption of 3/4 cup of cooked navy beans.
  Arms: Navy Beans (cooked)
Other: Red Kidney Beans (cooked) — One time consumption of 3/4 cup of cooked red kidney beans.
  Arms: Red Kidney Beans (cooked)
Other: Pinto Beans (cooked — One time consumption of 3/4 cup of cooked pinto beans.
  Arms: Pinto Beans (cooked)
Other: Black Beans (cooked) — One time consumption of 3/4 cup of cooked black beans.
  Arms: Black Beans (cooked)
Other: Lentils (cooked) — One time consumption of 3/4 cup of cooked lentils.
  Arms: Lentils (cooked)
Other: White Rice — One time consumption of 3/4 cup of cooked white rice.
  Arms: White Rice (cooked)

SUMMARY:
This is a single site, blinded, randomized, controlled study designed to examine phytochemical absorption, metabolism and excretion, as well as vascular health and satiety, after ingestion of 4 different bean varieties (pinto, navy, red kidney, black). Eligible participants will attend 6 in-person clinic visits for comparative testing of the 4 bean varieties versus lentils and rice.

DETAILED DESCRIPTION:
This is a single site, blinded, randomized, controlled study designed to examine phytochemical absorption, metabolism and excretion, as well as vascular health and satiety, after ingestion of 4 different bean varieties (pinto, navy, red kidney, black).

Recruitment will consist of a total of 8 volunteers. Volunteers will be recruited through advertisement from the local community.

The study will be conducted at the I.H. Asper Clinical Research Institute,located at the St. Boniface Hospital. Participants will be asked to provide written informed consent prior to participation in the study. Participants who have provided written consent will be asked to attend an in-patient visit to provide a fasting blood sample. Should the participant be eligible to participate, they will be scheduled for six study visits to assess the bioavailability, metabolism and excretion of phytochemicals present in beans compared to lentils and white rice.

Uptake, metabolism and excretion of phytochemicals present in different varieties of beans during acute phase testing in healthy individuals will be examined. Possible relationships between phytochemical composition of the beans, arterial function and satiety will be investigated as the secondary objective.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥18 and ≤50 years;
2. Normal blood lipid profile, creatinine ≥7 units/L and ≤56 units/L, alanine aminotransferase (ALT) ≥0.7 mg/dL and ≤1.3 mg/dL for men and ≥0.6 mg/dL and ≤1.1 mg/dL for women, and glycated hemoglobin <6%;
3. Blood pressure <140/90
4. Body mass index (BMI) ≥20 and <30;
5. Stable regime for the past 3 months if taking vitamin and mineral/dietary/ herbal supplements;
6. Agree not to eat beans or bean-based foods, lentils or lentil-based foods, or consume isoflavone supplements while participating in this study;
7. Willing to comply with the protocol requirements;
8. Willing to provide informed consent.

Exclusion Criteria:

1. Allergies to beans, bean flour or bean products, lentils or rice;
2. Presence of a clinically diagnosed disease affecting the circulatory, respiratory, immune, skeletal, urinary, muscular, endocrine, digestive, nervous or reproductive system that requires medical treatment;
3. Taking any prescribed medication in the last 3 months (with the exception of birth control) or supplements that affect gastrointestinal function in the last 3 months;
4. Weight loss of ≥3 kg of body weight within the 6 months prior to enrolling in the study;
5. Current (within the last month) bacterial, viral or fungal infection, or over-the-counter medication within the past 72 hours;
6. Pregnant or lactating;
7. Unable to obtain blood samples at the screening visit or the first study visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Composite measure of Absorption, Metabolism and Excretion of Phytochemicals | Timepoint 0 (prior to consumption), 0.5, 1.0, 1.5, 2, 4 and 6 hours post consumption
  Blood and urine samples will be analyzed using a differential analysis for metabolites (p<0.01 and fold changes ≥ 2) which will be achieved via principle component analysis (PCA), and partial least square (PLS).

SECONDARY OUTCOMES:
Changes in parameters of arterial stiffness through pulse wave analysis (PWA) | Time points 0 (prior to consumption) and 2 and 6 hours post consumption.
  A measure of changes in arterial stiffness as assessed via pulse wave analysis (PWA) using a Mobil-O-Graph PWA Monitor prior to consumption, at 2 hours and 6 hours post-consumption.
Satiety Questionnaire | 5 hours after consumption of study product
  Participants will complete a Satiety Questionnaire 5 hours after consumption of the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zahradka, PhD, Principal Investigator — University of Manitoba
Locations (1):
- St.Boniface Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Hanson MG, Zahradka P, Taylor CG. Lentil-based diets attenuate hypertension and large-artery remodelling in spontaneously hypertensive rats. Br J Nutr. 2014 Feb;111(4):690-8. doi: 10.1017/S0007114513002997. Epub 2013 Sep 24. PMID 24063808
- [Background] Zahradka P, Wright B, Weighell W, Blewett H, Baldwin A, O K, Guzman RP, Taylor CG. Daily non-soy legume consumption reverses vascular impairment due to peripheral artery disease. Atherosclerosis. 2013 Oct;230(2):310-4. doi: 10.1016/j.atherosclerosis.2013.07.048. Epub 2013 Aug 6. PMID 24075762
- [Background] Vinaixa M, Samino S, Saez I, Duran J, Guinovart JJ, Yanes O. A Guideline to Univariate Statistical Analysis for LC/MS-Based Untargeted Metabolomics-Derived Data. Metabolites. 2012 Oct 18;2(4):775-95. doi: 10.3390/metabo2040775. PMID 24957762
- [Background] Nyamundanda G, Gormley IC, Fan Y, Gallagher WM, Brennan L. MetSizeR: selecting the optimal sample size for metabolomic studies using an analysis based approach. BMC Bioinformatics. 2013 Nov 21;14:338. doi: 10.1186/1471-2105-14-338. PMID 24261687
- See also: Canadian Centre for Agri-Food Research in Health and Medicine — http://www.ccarm.ca